CLINICAL TRIAL: NCT02872064
Title: A Phase I/IIa, Open Label, Single Site Light Dose Escalation Trial of Single Dose Verteporfin Photodynamic Therapy (PDT) in Primary Breast Cancer
Brief Title: Treatment of Primary Breast Cancer Using PDT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09/0286
Record Dates: First submitted 2016-08-15; First posted 2016-08-18 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-03

CONDITIONS: Breast Neoplasms
Keywords: Early breast cancer; Photodynamic therapy; PDT; Visudyne; Verteporfin
MeSH Terms: conditions — Breast Neoplasms | interventions — Verteporfin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment with PDT (Experimental): A single intravenous injection of Verteporfin (0.4mg/kg) will be administered, at least 60minutes and up to 90 minutes before laser activation. A 690nm red laser light will be delivered with a diffuser laser fibre inserted through the skin into the breast tissue, with light dose escalation after every three patients. All patients will have fixed dose of the photosensitizer but variable light dose.
  Interventions: Drug: Verteporfin

INTERVENTIONS:
Drug: Verteporfin — Verteporfin (which is marketed under the brand name Visudyne) is the photosensitizer. Verteporfin is a benzoporphyrin derivative which is clinically active when formulated with liposomes. By itself the clinically recommended dose of Verteporfin is not cytotoxic. It produces cytotoxic agents only when activated by light in the presence of oxygen. When energy absorbed by the porphyrin is transferred to oxygen, highly reactive short lived singlet oxygen is generated. Singlet oxygen causes damage to biological structures, leading to local vascular occlusion, cell damage and cell death.
  Other Names: Visudyne

SUMMARY:
Phase I/IIA, open label, non-randomised, single site trial in patients with primary breast cancer.

DETAILED DESCRIPTION:
This is a phase I / IIa study recruiting patients diagnosed with primary breast cancer. Patients who have chosen mastectomy or wide local excision as their surgical option will be included. Patients will have a pre therapy MRI followed by photodynamic therapy. PDT involves intravenously injecting the photosensitizer Verteporfin (Visudyne) drug. This drug makes the tumour sensitive to light. A non-thermal light will then be shone in the tumour which brings about tissue necrosis (destruction). Although the drug dose will remain the same, the light dose will be escalated depending on patient response in accordance to a predefined algorithm (see section) to achieve a zone of necrosis of 12mm or a plateau of necrosis with incremental increase in light dose. An MRI will be performed immediately prior to the scheduled surgery. Pre and post PDT MRI changes will be correlated with the histological findings on the excised breast specimen. Should the minimum light dose for 12mm necrosis be established recruitment will continue until 12 patients have received this dose. These 12 patients will provide sample data on the size of tumour and area of necrosis detected by MRI and histology to enable sample size (power) calculations for future studies of PDT in primary breast cancer. This is a dose escalation study involving a minimum of twelve and a maximum of forty patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 30 or over
2. A uni-focal invasive ductal breast carcinoma or discrete uni-focal site which is deemed suitable for PDT within a multifocal invasive ductal carcinoma in a single breast.
3. Patients who have opted for mastectomy or wide local excision as primary treatment.
4. Capable of giving written informed consent

Exclusion Criteria:

1. Patients who are not undergoing surgery as their primary treatment.
2. Patients undergoing surgery for DCIS without invasive breast cancer.
3. Patients with Lobular cancer
4. Patients with Necrotic tumours
5. Distant metastatic disease.
6. Patients will be excluded if they have porphyria or are sensitive to verteporfin (visudyne).
7. Patients who have severe cardiovascular disease.
8. Patients with severe or uncontrolled systemic disease e.g. hepatic impairment.
9. Patients with laboratory findings that make it undesirable for the patient to participate in the trial.
10. Male breast cancer patients
11. Pregnancy and lactation.
12. No patients with any psychiatric disorder making reliable informed consent impossible.
13. Patients will be excluded if taking part in any other trial of an experimental medicine
14. Patients will be excluded if taking endocrine therapy drugs that could confound the results.

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Establish the minimum effective light dose | One month
  To establish the minimum light dose, in the range 20Joules/ (cm of light diffuser length) but not exceeding 90J/cm, required to induce an area of necrosis with a diameter of at least 12mm in line perpendicular to the fibre on microscopic examination or to achieve a plateau with no increasing necrosis as the light dose increases.

SECONDARY OUTCOMES:
Compare final histology with post PDT MRI. | One month
  To assess the response of the Photodynamic Therapy on primary breast cancer via radiology using pre and post PDT MRI and comparing this with final histology. Measurements will be made of the diameter of necrosis on MRI scan which will be correlated with the histological measurement.
Assess affect of PDT on normal breast tissue. | One month
  To look at the effect of Photodynamic Therapy on the abnormal breast tissue and study if necrosis extends to normal breast tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Mo RS Keshtgar, Principal Investigator — Royal Free NHS Trust
Locations (1):
- Royal Free Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All requests for data sharing will adhere to the UCL Surgical & Interventional Trials Unit (SITU) data sharing agreement policy. UCL Medical School is supportive of data sharing and will endeavour to assist in requests for data sharing. These data will be held at UCL on secure servers and will not be released to any third parties until the final study report has been published. All requests for access to the data will be formally requested through the use of a SITU data request form which will state the purpose, analysis and publication plans together with the named collaborators. All requests are dealt with on a case by case basis. All requests will be logged and those successful will have a data transfer agreement which will specify appropriate acknowledgement of the Royal Free Hospital, the sponsor, and funders.